CLINICAL TRIAL: NCT00781742
Title: A Phase IIb, Multicenter, Randomized, Double-blind, Parallel Group, Placebo-controlled Efficacy and Safety Study of Adjunctive AZD6765 in Subjects With Severe Major Depressive Disorder (MDD) and a History of Poor Response to Antidepressants
Brief Title: AZD6765 Severe Major Depressive Disorder (MDD) IV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D6702C00009
Record Dates: First submitted 2008-10-27; First posted 2008-10-29 (Estimated); Last update posted 2012-07-25 (Estimated); Status verified 2012-07

CONDITIONS: Major Depressive Disorder
Keywords: Depression; Depressive Disorder; MDD
MeSH Terms: conditions — Depressive Disorder, Major; Depression; Depressive Disorder | interventions — AZD6765

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- 1 (Experimental): 100 mg iv once per dosing day
  Interventions: Drug: AZD6765
- 2 (Experimental): 150 mg iv once per dosing day
  Interventions: Drug: AZD6765
- 3 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD6765 — IV once per dosing day, multiple times during the treatment period
  Arms: 1; 2
Drug: Placebo — 0.9% saline IV once per dosing day multiple times during the treatment period
  Arms: 3

SUMMARY:
The purpose of this research study is to determine whether AZD6765 has an effect on the patient's depression when taken together with current depression medication. In addition, information will be gathered on how well AZD6765 is tolerated, investigate the levels of AZD6765 and the levels of the current depression medication in the blood. In addition, the research staff will determine if AZD6765 has any mood or calming effects (how you feel).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent before any study-related procedures start.
* The patient is previously diagnosed with Major Depressive Disorder (MDD) and currently taking an antidepressant for at least 6 weeks.
* Patient has a history of poor response to 1 or more antidepressants (in addition to the antidepressant the patient is taking at enrollment) after exposure at adequate doses or maximum tolerated doses for ≥4 weeks.

Exclusion Criteria:

* Patient has a lifetime history of schizophrenia, bipolar, psychosis or psychotic depression.
* Patient has a lifetime history of failure to ECT therapy.
* Patient is pregnant or breast feeding.
* Length of current episode of depression exceeds ≥2 years.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2008-10; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
To give evidence of an antidepressant effect versus placebo, given together with another antidepressant confirmed by change in the MADRS total score | Baseline to week 3

SECONDARY OUTCOMES:
To determine if the antidepressant effect can be achieved at week 3 with AZD6765 (100 or 150 mg/infusion) versus placebo by assessing a change from baseline to week 3 in the MADRS total score. | 3 weeks
To evaluate the rapid antidepressant efficacy of AZD6765 at 1 day after a first infusion, as assessed by a change in the Quick Inventory of Depressive Symptomology Self-Report 16-item scale (QIDS-SR-16) total score. | baseline to Day 1
• To assess the safety and tolerability of multiple infusions when administered concomitantly with other anti-depressants by incidence of AEs. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael Castiglione, Study Director — AstraZeneca; Gerard Sanacora, Principal Investigator — Yale University
Locations (27):
- United States (27):
  - Research Site, Little Rock, Arkansas
  - Research Site, Los Angeles, California
  - Research Site, Orange, California
  - Research Site, San Diego, California
  - Research Site, Santa Ana, California
  - Research Site, Hartford, Connecticut
  - Research Site, New Haven, Connecticut
  - Research Site, Boca Raton, Florida
  - Research Site, Gainsville, Florida
  - Research Site, Hollywood, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Roswell, Georgia
  - Research Site, Hoffman Estates, Illinois
  - Research Site, Joliet, Illinois
  - Research Site, Overland Park, Kansas
  - Research Site, Lake Charles, Louisiana
  - Research Site, Shreveport, Louisiana
  - Research Site, Haverhill, Massachusetts
  - Research Site, St Louis, Missouri
  - Research Site, Willingboro, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, Rochester, New York
  - Research Site, East Stroudsburg, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas

REFERENCES:
- [Derived] Dean RL, Hurducas C, Hawton K, Spyridi S, Cowen PJ, Hollingsworth S, Marquardt T, Barnes A, Smith R, McShane R, Turner EH, Cipriani A. Ketamine and other glutamate receptor modulators for depression in adults with unipolar major depressive disorder. Cochrane Database Syst Rev. 2021 Sep 12;9(9):CD011612. doi: 10.1002/14651858.CD011612.pub3. PMID 34510411
- [Derived] Sanacora G, Smith MA, Pathak S, Su HL, Boeijinga PH, McCarthy DJ, Quirk MC. Lanicemine: a low-trapping NMDA channel blocker produces sustained antidepressant efficacy with minimal psychotomimetic adverse effects. Mol Psychiatry. 2014 Sep;19(9):978-85. doi: 10.1038/mp.2013.130. Epub 2013 Oct 15. PMID 24126931